CLINICAL TRIAL: NCT01566097
Title: Development and Application of Culturally-Appropriate Decision Aids for Smoking Cessation in Korea: a Single Arm Intervention Trial With Historical Control
Brief Title: Intervention Trial of Culturally-Appropriate Decision Aids for Smoking Cessation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Dong Wook Shin, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-1202-032-397
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Cigarette Smoking; Tobacco Use Disorder; Nicotine Dependence; Smoking Cessation
Keywords: Cluster randomized trial; Decision aids; Culturally-appropriate decision aids
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): This study is cluster randomized trial, and the randomization level is physician. Current smokers seen by physician allocated into intervention group were provided with Smoking Cessation Decision Aids along with study questionnaires. The intervention was Smoking Cessation Decision Aids provided to current smokers.
  Interventions: Device: Smoking Cessation Decision Aids
- Control group (No Intervention): Current smokers seen by physician allocated into control group were provided with only study questionnaires and usual care.

INTERVENTIONS:
Device: Smoking Cessation Decision Aids — The decision aids were developed through: 1) literature review; 2) qualitative interviews with Korean smokers from various backgrounds; 3) expert opinions. They were in the form of short educational videos (flash), displayed by Apple's iPad.
  The decision aids contained the followings, in proper Korean social and cultural context:
  1. Information on the risk of continued smoking and benefits of cessation
  2. Messages that address common misbeliefs regarding smoking cessation services and medications
  3. Information on possible smoking cessation options, their efficacy, side effects, costs, etc.
  The choices given in the decisions aid were:
  1. Behavioral only
  2. Nicotine replacement therapy
  3. Bupropion
  4. Varenicline
  Arms: Intervention group

SUMMARY:
Despite the establishment of various smoking cessation methods, including pharmacological intervention, only a small proportion of smokers who visit doctors choose to receive such assistance. Such under-utilization is especially apparent in some cultures, as in the case of Korea, where a government survey showed that only 0.5% of current or formal smoker reported they had been prescribed smoking cessation medication. Shame in asking for help for an addictive disorder has been recognized as one of the most recognized cultural barrier in Asian-American population. It is clear that culturally focused studies on smoking cessation is warranted.

Patient decision aids are tools that help people become involved in decision making by providing information about the options and outcomes and by clarifying personal values. Patient decision aids have been developed to help patients decide whether to quit smoking or not, or whether to use smoking medication or not. However, such previous studies have only been focused on western populations.

The main purpose of this study is to develop a culturally appropriate decision aid for smoking cessation for the Korean population, as well as evaluate its effect on their decision to use smoking cessation medication. The investigators expect that culturally tailored smoking cessation decision aids would increase knowledge about efficacy of smoking cessation, make people have more positive attitudes toward smoking cessation medication, encourage people to discuss about smoking cessation medication with their physicians. Ultimately the investigators expect it would increase usage of smoking cessation medication and enhance the quitting rate of smoking, which is a very important clinical issue.

DETAILED DESCRIPTION:
Reluctance to use smoking cessation medication has been identified as most important barriers to successful smoking cessation in the general population. While pharmacologic intervention, especially prescription drug, is recommended by the guideline as most effective therapy for smoking cessation, only a few smokers who visit doctors take medication reflecting serious underutilization of the pharmacologic intervention. Although it seems to be at least equally effective in Asian population compared with the Western counterpart (Fagerstrom, 2010), data from Korean National Health and Nutrition Examination Survey shows that only 0.5% of current or formal smoker reported they had been prescribed smoking cessation medication, far less than those reported from US, UK, Australia, and Canada.

Culture might also affect the treatment-seeking behavior related to smoking cessation. Data from the tobacco helpline in California showed that about 40 percent of the Asian callers to the tobacco helpline were friends or family members compared to six percent of the calls for non-Asian (Zhu SH, 2002). This suggests that Asian Americans and Pacific Islanders may be less likely to ask for help for themselves or that family members are more likely to ask for help for their loved one. This implicates the need to involve family members in treatment from the very beginning, which is a different concept than that seen in the themes of self reliance and personal responsibility among Western cultures (Fong, 2007). In general, it is recognized that Asian Americans with addictive disorders face several cultural and practical barriers to treatment and the result has been an underutilization of addiction and mental health treatment. For example, shame in asking for help for an addictive disorder is recognized as one of the most recognized cultural barrier in this population (Fong, 2007). A few preliminary interventions were targeted to Asian Americans (for example, Suc Khoe La Vang for Vietnamese American and Lay-led smoking cessation approach for South East Asian men, etc), and provided some preliminary evidence for the effectiveness of such culturally-appropriate smoking cessation intervention (Chen, 2001).

To our knowledge, no research has focused on the cultural aspect of smoking cessation in Korean smokers. Asian's general reluctance to use mental health services, fear of stigma of lack of willpower, family issues might be some hypothesized examples of culture-specific barriers to medication use, in addition to more universal barriers like lack of knowledge of possible treatment options and their efficacy and fear of side effects. Understanding the Korean smoker's perspectives on the way of smoking cessation might be a key to the development of effective smoking cessation intervention in this population. However, there is a lack of detailed research on the Korean smokers' cultural beliefs and attitudes toward the smoking cessation, especially the use of smoking cessation medication.

Patient decision aids are tools that help people become involved in decision making by providing information about the options and outcomes and by clarifying personal values. It promotes shared decision making between the patient and practitioner, saves physician's time, and reduces practice variation. In smoking cessation area, patient decision aids has been developed to help the patients decide on whether to quit smoking or not (NHS, UK), and on whether to use smoking cessation medication or not (Healthwire, US; Willemsen, 2006). However, those decision aids were targeted to the Western population, thus limiting the generalizability of the utility of such tools in the population from other culture. To our best knowledge, there is no decision aid specifically tailored for Korean smokers, and we would like to develop one and evaluate its effect on their decision to use smoking cessation medication through this study.

The primary objectives of this study are: 1) to determine the effectiveness of culturally-tailored smoking cessation decision aids by comparing the proportion of using smoking cessation medication in Korean smokers visiting primary care clinic and health screening center with control, and 2) to identify the factors associated with the decision to use the smoking cessation medication, including sociodemographic, medical, behavioral and cognitive factors, etc. The secondary objective of this study is to determine the smoking cessation rates and use of smoking cessation medication in real world setting and identify the factors associated with smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* being age 18 years or older
* having smoked at least one puff in past 7 days

Exclusion Criteria:

* current enrollment in other substance abuse treatment program
* being pregnant
* being unable to communicate in Korean

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-02 (Actual); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of Smokers Who Are Prescribed Smoking Cessation Medication | 1 month after viewing decision aids
  Patients who visited primary care clinic and health screening center were to be targeted for recruitment of the study. Current smokers seen by physician allocated into intervention group were provided with Smoking Cessation Decision Aids. The proportion of smokers who are prescribed smoking cessation medication within 1 month after reading Decision Aids will be compared with that of control group. The information will be recruited from medical chart.

SECONDARY OUTCOMES:
Abstinence Rate (Point Prevalence) | 6 months after viewing decision aids
  Participants are assessed for their abstinence rate according to their choices via telephone interview, as the final outcome of the study. The abstinence rate of patients in intervention arm will be compared with that of control arm
Proportion of Smokers Who Are Prescribed Smoking Cessation Medication | 6 month after viewing decision aids
  Participants are expected to choose from various treatment choices after initially viewing the decision aids, from no treatment to smoking cessation medication. Proportion of smokers who are prescribed smoking cessation medication within 6 months after reading Decision Aids will be compared with that of control group. The information are assessed via telephone interview.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wook Shin, MD,MBA,DrPH, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Result] Buck D, Morgan A. Smoking and quitting with the aid of nicotine replacement therapies in the English adult population. Results from the Health Education Monitoring Survey 1995. Eur J Public Health. 2001 Jun;11(2):211-7. doi: 10.1093/eurpub/11.2.211. PMID 11420814
- [Result] Willemsen MC, Wiebing M, van Emst A, Zeeman G. Helping smokers to decide on the use of efficacious smoking cessation methods: a randomized controlled trial of a decision aid. Addiction. 2006 Mar;101(3):441-9. doi: 10.1111/j.1360-0443.2006.01349.x. PMID 16499517